CLINICAL TRIAL: NCT03407118
Title: Pharmacokinetics and Glucodynamics of LY900014 Compared to Insulin Lispro (Humalog) Following Single Dose Administration in Japanese Patients With Type 1 Diabetes Mellitus
Brief Title: A Study of LY900014 in Japanese Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16645; I8B-MC-ITRZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Results first posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY900014 (Experimental): Single, 15 units (U)LY900014 administered subcutaneously (SC) in one of two study periods in Japanese Patients With Type 1 Diabetes Mellitus (T1DM).
  Interventions: Drug: LY900014
- Insulin Lispro (Humalog) (Active Comparator): Single, 15 U insulin lispro administered SC in one of two study periods in Japanese Patients With Type 1 Diabetes Mellitus.
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900014 — Administered SC.
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin Lispro — Administered SC.
  Other Names: LY275585; Humalog
  Arms: Insulin Lispro (Humalog)

SUMMARY:
This study will compare LY900014, a drug that lowers blood sugar, with insulin lispro (Humalog). Both drugs will be given by injection under the skin of the abdomen. This study will be conducted in participants with type 1 diabetes to investigate how quickly and how much LY900014 is absorbed and the effect of LY900014 on blood sugar levels in comparison with insulin lispro. The study will last about 3 to 6 weeks for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are Japanese male or female participant with a diagnosis of T1DM, based on the World Health Organization classification, for at least 1 year prior to screening
* Have a body mass index (BMI) of 18.5 to 30.0 kilograms per square meter (kg/m²)
* Have a glycated hemoglobin <9.0% at screening

Exclusion Criteria:

* Have, except for current regimen of insulin therapy and concomitant medication(s), regular use of or intended use of any over-the-counter or prescription medications or nutritional supplements that treat hyperglycemia or insulin resistance or that promote weight loss within 14 days before dosing
* Are receiving chronic (lasting longer than 14 consecutive days) systemic or inhaled glucocorticoid therapy (excluding topical, intra-articular, and intraocular preparations), or have received such therapy within the 4 weeks before screening
* Have a history of renal impairment (exclusion only if estimated glomerular filtration rate [GFR] <60 milliliters/minute/1.73 square meters [GFR is estimated according to a formula recommended by the Japanese Society of Nephrology]), or have a serum creatinine level ≥126 micromoles per liter (μmol/L) (>1.42 milligrams per deciliter [mg/dL]) (male) or ≥111 μmol/L (>1.25 mg/dL) (female)
* Have a history of deep vein thrombosis of the leg, or repeated episodes of deep leg vein thrombosis in first-degree relatives (parents, siblings, or children), as determined by the investigator
* Have proliferative retinopathy or maculopathy and/or severe neuropathy; in particular, autonomic neuropathy, as determined by the investigator based on a recent (<1.5 years) ophthalmologic examination
* Have had any significant changes in insulin regimen and/or unstable blood glucose control within the past 3 months prior to screening, as determined by the investigator
* Require daily insulin treatment >1.5 units per kilogram (U/kg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-02-17 (Actual); Primary Completion 2018-06-23 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- LY900014\Insulin Lispro (Humalog): Period 1: A single dose of 15 Units (U) LY900014 administered subcutaneously (SC) .
  Period 2: A single dose of 15 U insulin lispro (Humalog) administered SC with up to 28 days between doses
- Insulin Lispro (Humalog)\LY900014: Period 1: A single dose of 15 U insulin lispro (Humalog) administered SC.
  Period 2: A single dose of 15 Units (U) LY900014 administered subcutaneously (SC) . with up to 28 days between doses.
Period: Period 1
Arm/Group | LY900014\Insulin Lispro (Humalog) | Insulin Lispro (Humalog)\LY900014
Started | 14 | 17
Received at Least 1 Dose of Study Drug | 14 | 17
Completed | 14 | 17
Not Completed | 0 | 0
Period: Period 2
Arm/Group | LY900014\Insulin Lispro (Humalog) | Insulin Lispro (Humalog)\LY900014
Started | 14 | 17
Received at Least 1 Dose of Study Drug | 13 | 17
Completed | 13 | 17
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- All Participants: All randomized participants who received at least 1 dose of study drug.
Arm/Group | All Participants
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 31
Weight [Mean (Standard Deviation); unit: kilograms] | 59.62 (8.29)
Height [Mean (Standard Deviation); unit: centimeters] | 161.35 (7.44)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per meter squared] | 22.85 (2.44)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro Area Under the Concentration Curve Zero to 10 Hours (AUC 0-10h) Following Administration of Each Treatment Arm
Description: PK: Insulin Lispro AUC from time zero to 10 hours
Time Frame: Predose, 5 minutes (min), 10 min, 15 min, 20 min, 25 min, 30 min, 35 min, 40 min, 45 min, 50 min, 55 min, 60 min, 70 min, 90 min, 120 min, 150 min, 180 min, 240 min, 300 min, 360 min, 420 min, 480 min, 540 min, and 600 min postdose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomols times hour per Liter
Groups:
- 15 U LY900014: A single dose of 15 Units (U) LY900014 administered subcutaneously (SC) in one of two study periods.
- 15 U Insulin Lispro (Humalog): A single dose of 15 U insulin lispro (Humalog) administered SC in one of two study periods.
Arm/Group | 15 U LY900014 | 15 U Insulin Lispro (Humalog)
Number analyzed (Participants) | 31 | 30
picomols times hour per Liter | 1930 (59) | 1980 (20)
Statistical Analysis 1: Comparison: 15 U LY900014 vs 15 U Insulin Lispro (Humalog); Test type: Superiority; ratio of least square means = 0.967, 95% CI 2-sided [0.803 to 1.17]

2. Secondary Outcome: Glucodynamics (GD): Total Amount of Glucose Infused (Gtot) Over Duration of Clamp Following Administration of Each Treatment Arm
Description: Gtot Over Duration of Clamp for Each Treatment Arm. Gtot is the total glucose infusion over the clamp duration (10 hours) and is used to measure the study drug action over time as measured by the euglycemic clamp (EC) procedure. During the euglycemic clamp procedure, blood glucose concentrations are held constant after the administration of study treatment by adjusting the exogenous glucose infusion rate.
Time Frame: Predose, every minute from run-in and for the duration of the EC until up to 10 hours postdose
Population: All randomized participants who received at least 1 dose of study drug and had evaluable GD data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams per kilogram
Arm/Group | 15 U LY900014 | 15 U Insulin Lispro (Humalog)
Number analyzed (Participants) | 31 | 30
milligrams per kilogram | 1190 (54) | 1250 (34)

ADVERSE EVENTS:
Time Frame: Baseline up to 56 weeks
Description: All randomized participants.
Groups:
- LY900014: A single dose of 15 Units (U) LY900014 administered subcutaneously (SC) . in one of two study periods.
- Insulin Lispro (Humalog): A single dose of 15 U insulin lispro (Humalog) administered SC in one of two study periods.
Arm/Group | LY900014 | Insulin Lispro (Humalog)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 6/31 | 7/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY900014 (N=31) | Insulin Lispro (Humalog) (N=30)
nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT03407118/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT03407118/SAP_001.pdf